CLINICAL TRIAL: NCT00924885
Title: Experience of Pain During Oocyte Retrieval- a Comparison Between Two Aspiration Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vitrolife-needle-01
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Infertility
Keywords: Reproductive Medicine; Fertilization in Vitro; Oocyte retrieval; Local anaesthesia; Aspiration needle
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thin Follicle Aspiration Needle (Experimental): Transvaginal oocyte retrieval was performed under local anaesthesia and under guidance of ultrasound with the RN needle that had an outer diameter of 0.9 mm (20 gauge) and inner diameter of 0.6 mm for the last 50 mm from the tip of the needle and an outer diameter of 1.4 mm (17 gauge) and inner diameter of 1 mm for the remaining length of the needle. The puncture procedure was performed according to each clinic's standard routine. Aspiration pressure was kept at a negative pressure between 90 and 120 mmHg.
  Interventions: Device: Swemed Follicle Aspiration Set Reduced Single Lumen
- Standard Follicle Aspiration Needle (Active Comparator): Transvaginal oocyte retrieval was performed under local anaesthesia and under guidance of ultrasound with the SN needle that had an outer diameter of 1.4 mm (17 gauge) and inner diameter of 1 mm for the remaining length of the needle. or the SN with an outer diameter of 1.4 mm (17 gauge) and inner diameter of 1 mm for the whole length of the needle.
  The puncture procedure was performed according to each clinic's standard routine. Aspiration pressure was kept at a negative pressure between 90 and 120 mmHg.
  Interventions: Device: Swemed Follicle Aspiration Set Single Lumen (1.4 mm)

INTERVENTIONS:
Device: Swemed Follicle Aspiration Set Reduced Single Lumen — Thin tip to penetrate the tissue
  Arms: Thin Follicle Aspiration Needle
Device: Swemed Follicle Aspiration Set Single Lumen (1.4 mm) — Standard (1.4 mm) needle to penetrate the tissue
  Arms: Standard Follicle Aspiration Needle

SUMMARY:
The purpose of the study is to compare the pain experience between the patients that have had their transvaginal oocytes retrieval with ultrasound guidance performed with reduced single lumen needle (Vitrolife Sweden AB, Gothenburg) with the patients that have had follicle aspiration needle, 1.4 outer diameter (Vitrolife Sweden AB, Gothenburg), during the procedure.

DETAILED DESCRIPTION:
Although the patient is sedated and local analgesia has been given, transvaginal oocytes retrieval with ultrasound guidance can still cause a lot of pain, both during and after the procedure. To reduce the pain, some clinics prefer to use needles as thin as 0.8 mm (outer diameter, OD). A disadvantage with these needles is the increased aspiration time. Therefore a new needle has been developed that has the possibility to reduce pain without a large increase in aspiration time. The needle has a 50 mm long tip with an outer diameter of 0.9 mm. The remaining part of the needle is 300 mm long with an outer diameter of 1.4 mm.

ELIGIBILITY:
Inclusion Criteria:

* The patient has signed an informed consent form before the oocyte retrieval
* The patient is undergoing oocyte retrieval with local anaesthesia
* The patient can speak and understand Swedish

Exclusion Criteria:

* The patient has previously participated in Vitrolife-needle-01 study
* The patient has a body mass index ≥35
* Other contra indicator for oocyte retrieval

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Hillensjö, MD PhD, Principal Investigator — Fertility Center Scandinavia
Locations (4):
- Sweden (4):
  - IVF-kliniken Falun, Falun
  - Fertilitetscentrum Göteborg, Gothenburg
  - Reproduktionmedicinskt Center, Universitetssjukhuset MAS, Malmo
  - Fertilitetsenheten K59 Karolinska Universitetssjukhuset, Huddinge, Stockholm

REFERENCES:
- [Derived] Wikland M, Blad S, Bungum L, Hillensjo T, Karlstrom PO, Nilsson S. A randomized controlled study comparing pain experience between a newly designed needle with a thin tip and a standard needle for oocyte aspiration. Hum Reprod. 2011 Jun;26(6):1377-83. doi: 10.1093/humrep/der100. Epub 2011 Apr 5. PMID 21467200
- See also: Link to the published article — http://www.ncbi.nlm.nih.gov/pubmed/21467200

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thin Follicle Aspiration Needle | Standard Follicle Aspiration Needle
Started | 129 | 128
Completed | 126 | 124
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thin Follicle Aspiration Needle | Standard Follicle Aspiration Needle | Total
Number analyzed (Participants) | 129 | 128 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 129 | 128 | 257
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (4.7) | 34.4 (4.2) | 34.3 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 128 | 257
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 129 | 128 | 257

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale
Description: Rating of pain was performed by self-assessment by means of Visual Analogue Scale (VAS) consisting of a line oriented vertically on a paper with a range from 0 mm (no pain) to 100 mm (unbearable pain).
Time Frame: After the oocyte retrieval and before the patient leaves the operation room e.g. within a maximum of 30 minutes.
Measure: Mean (Standard Deviation); unit: 0-100 mm
Arm/Group | Thin Follicle Aspiration Needle | Standard Follicle Aspiration Needle
Number analyzed (Participants) | 126 | 124
0-100 mm | 21.0 (17.5) | 26.0 (19.9)
Statistical Analysis 1: Comparison: Thin Follicle Aspiration Needle vs Standard Follicle Aspiration Needle; The primary end-point was the 'overall pain experience', evaluated as described previously. Assuming the mean overall pain in the RN group to be 27 mm (value chosen after analysis of data from a previous study, Cerne et al., 2006) on VAS, with a standard deviation (SD) of 21.5 mm, 121 patients in each group would be needed to demonstrate a decrease in overall pain of 8 mm (30%) with 80% power and a significance level of 0.05 (two-tailed tests); Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Intervention Because of Bleeding
Description: Vaginal bleeding during or after the procedure was graded subjectively by the physician as (i) less than normal, (ii) normal or (iii) more than normal.
Time Frame: During and directly after oocyte retrieval
Population: Bleeding during follicle aspiration was graded in all patients included in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Follicle Aspiration Needle: Transvaginal oocyte retrieval was performed under local anaesthesia and under guidance of ultrasound with the SN needle that had an outer diameter of 1.4 mm (17 gauge) and inner diameter of 1 mm for the remaining length of the needle. or the SN with an outer diameter of 1.4 mm (17 gauge) and inner diameter of 1 mm for the whole length of the needle.
  The puncture procedure was performed according to each clinic's standard routine. Aspiration pressure was kept at a negative pressure between 90 and 120 mmHg.
  Swemed Follicle Aspiration Set Single Lumen (1.4 mm): Standard (1.4 mm) needle to penetrate the tissue
Arm/Group | Thin Follicle Aspiration Needle | Standard Follicle Aspiration Needle
Number analyzed (Participants) | 126 | 124
Participants
  Less than normal bleeding | 40 | 24
  Normal bleeding | 80 | 93
  Bleeding more than normal | 6 | 7

ADVERSE EVENTS:
Time Frame: Records of serious events were collected over a period of one week after oocyte pick-up (OPU)
Description: Definitions same as used by .gov
Arm/Group | Thin Follicle Aspiration Needle | Standard Follicle Aspiration Needle
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/128
Other Adverse Events (participants affected / at risk) | 0/129 | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No